CLINICAL TRIAL: NCT01295944
Title: Phase II Trial of Carboplatin and Bevacizumab for the Treatment of Recurrent Low-Grade and Anaplastic Supratentorial, Infratentorial and Spinal Cord Ependymoma in Adults: A Multi-Center Trial
Brief Title: Carboplatin and Bevacizumab for Recurrent Ependymoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kevin Camphausen, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 160009; 16-C-0009
Record Dates: First submitted 2011-02-11; First posted 2011-02-15 (Estimated); Results first posted 2021-12-28 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Ependymoma; Anaplastic Ependymoma
Keywords: Chemotherapy; Brain Tumor; Spinal Cord Tumor; Malignancy; Neurologic
MeSH Terms: conditions — Ependymoma; Brain Neoplasms; Spinal Cord Neoplasms; Neoplasms; Neurologic Manifestations | interventions — Carboplatin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 1/Carboplatin and Bevacizumab for Recurrent Ependymoma (Experimental): The total duration of treatment will be 6 cycles. After cycle 6, carboplatin should be discontinued, but bevacizumab may be continued at the discretion of the treating physician.
  Interventions: Drug: Carboplatin; Drug: Bevacizumab

INTERVENTIONS:
Drug: Carboplatin — Carboplatin will be given on day 1 of each cycle; the carboplatin dose should be calculated using the Calvert formula: Carboplatin dose (mg) = target Area Under the Curve (AUC) x (Creatinine clearance (CrCl) + 25; The total duration of treatment will be 6 cycles. After cycle 6, carboplatin should be discontinued.
  Other Names: Paraplatin
Drug: Bevacizumab — Bevacizumab will be administered on days 1 and 15 of each cycle. Bevacizumab will be administered at a dose of 10 mg/kg; The total duration of treatment will be 6 cycles. After cycle 6, bevacizumab may be continued at the discretion of the treating physician.
  Other Names: Avastin

SUMMARY:
The goal of this clinical research study is to learn if the combination of bevacizumab and carboplatin can help to control recurrent ependymoma. The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
Background:

* Ependymomas are glial based tumors arising from the ependymal lining of the ventricular system and central canal of the spinal cord
* These tumors affect both adults and children and represent approximately 1.2%-7.8% of all intracranial cancers.
* Currently, the standard therapy for newly diagnosed low-grade ependymoma includes total surgical excision, when possible, followed by radiation therapy. Complete surgical resection is often not possible because of the location of the tumor and the concern for damage to surrounding eloquent brain during surgery. The situation is even more critical for patients with anaplastic ependymomas because of the higher proliferative rate and greater propensity for tumor infiltration into surrounding normal brain, preventing any possibility of complete tumor removal by surgery.
* For patients with the more aggressive anaplastic ependymoma, chemotherapy is often administered either before or after the radiation in the hope that infiltrating tumor cells will be eliminated.
* Extensive experience has been gathered with the use of bevacizumab in other neuroepithelial tumors such as malignant gliomas. Based on the interesting results observed in the reported small series of patients with recurrent ependymomas treated with bevacizumab, as well as on the evidence of vascular endothelial growth factor (VEGF)-promoted angiogenesis in these tumors, we designed a phase II study to test the efficacy of bevacizumab in patients with recurrent ependymoma. As results in most types of tumors have indicated that anti-angiogenesis therapies are more effective when given in combination with cytotoxic chemotherapy, in this study bevacizumab will be combined with carboplatin. The choice of carboplatin is justified by the fact that, as detailed above, this remains the most effective agent in this disease, and extensive toxicity data is available for the combination of bevacizumab and carboplatin in a variety of tumor types, including glioblastomas (GBMs).

Objective:

To evaluate the efficacy of carboplatin and bevacizumab for the treatment of recurrent low grade or anaplastic ependymoma. The primary endpoint will be progression-free survival (PFS) at one year.

Design:

* This is a phase II study to evaluate the efficacy of carboplatin and bevacizumab for the treatment of recurrent low grade or anaplastic ependymoma. This trial is designed utilizing a Simon optimal two-stage design.
* Carboplatin will be given on day 1 of each cycle. Bevacizumab will be administered on days 1 and 15 of each cycle. The total duration of treatment will be 6 cycles. After cycle 6, carboplatin should be discontinued, but bevacizumab may be continued at the discretion of the treating physician.
* Patients will be monitored for hematologic or serologic evidence of myelosuppression, hepatic injury, renal injury, and electrolyte disturbances and for clinical evidence of other toxicity.

ELIGIBILITY:
INCLUSION CRITERIA:

* Histologically proven intra-cranial or spinal ependymoma or anaplastic ependymoma. There must be pathologic or imaging confirmation of tumor progression or regrowth.
* The patient must have at least 1 block of tissue or 15 unstained slides at a minimum available for central pathology review and molecular profiling of the tissue sample.
* All patients must sign an informed consent indicating that they are aware of the investigational nature of this study. Patients must have signed an authorization for the release of their protected health information.
* Patients must be greater than or equal to 18 years old.
* Patients must have a Karnofsky performance status of > 60.
* Patients must have adequate bone marrow function (white blood cell (WBC) greater than or equal to 3,000/microliter, absolute neutrophil count (ANC) greater than or equal to 1,500/mm^3, platelet count of greater than to equal to 100,000/mm^3, and hemoglobin greater than or equal to 10 gm/dl), adequate liver function (Serum glutamic oxaloacetic transaminase (SGOT) [aspartate aminotransferase (AST) <92.5 Units/L] and bilirubin less than or equal to 1.5 mg/dL), and adequate renal function (creatinine < 1.5 mg/dL and calculated creatinine clearance greater than or equal to 60 cc/min) before starting therapy. Eligibility level for hemoglobin may be reached by transfusion.
* Patients must have shown unequivocal radiographic evidence for tumor progression by magnetic resonance imaging (MRI) or computed tomography (CT) scan.
* At the time of registration: Patients must have recovered from the toxic effects of prior therapy: greater than or equal to 28 days from any investigational agent, greater than or equal to 28 days from prior cytotoxic therapy, greater than or equal to 14 days from vincristine, greater than or equal to 42 days from nitrosoureas, greater than or equal to 21 days from procarbazine administration, and greater than or equal to 7 days for non-cytotoxic agents, e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid, etc. (radiosensitizer does not count). Any questions related to the definition of non-cytotoxic agents should be directed to the Principal Investigator.
* Patients having undergone recent resection of recurrent or progressive tumor will be eligible as long as all of the following conditions apply:
* They have recovered from the effects of surgery.
* A minimum of 28 days have elapsed from the day of surgery to the day of registration Step 2.
* For core or needle biopsy, a minimum of 7 days must have elapsed prior to registration Step 2.
* Residual disease following resection of recurrent ependymoma is not mandated for eligibility into the study. To best assess the extent of residual disease post-operatively, a CT/ MRI should be done no later than 96 hours in the immediate post-operative period or at least 4 weeks post-operatively, within 14 days prior to consent. If the within 96-hour after surgery scan is more than 14 days before consent the scan needs to be repeated. If the steroid dose is increased between the date of imaging and consent, a new baseline MRI/CT is required on a stable steroid dosage for at least 5 days.
* Patients must have failed prior radiation therapy* and must have an interval of greater than or equal to 42 days from the completion of radiation therapy to study entry. Note: Patients with an indication for craniospinal radiotherapy (i.e., extensive leptomeningeal disease) but have refused palliative craniospinal radiotherapy are eligible.
* Patients with prior therapy that included interstitial brachytherapy or stereotactic radiosurgery must have confirmation of true progressive disease rather than radiation necrosis based upon either positron emission tomography (PET) or Thallium scanning, MR spectroscopy, or surgical/pathological documentation of disease.
* Women of childbearing potential must have a negative B (Beta)-human chorionic gonadotropin (HCG) pregnancy test documented within 14 days prior to registration.
* Women of childbearing potential and male participants agree to practice adequate contraception.

EXCLUSION CRITERIA:

* Patients with any significant medical illnesses that in the investigators opinion cannot be adequately controlled with appropriate therapy or would compromise the patients ability to tolerate this therapy.
* Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma insitu of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years are ineligible.
* Patients with an active infection or serious intercurrent medical illness.
* Patients found to be pregnant/breast feeding. Patients must not be pregnant because animal studies show that carboplatin and bevacizumab are teratogenic
* Patients with any disease that will obscure toxicity or dangerously alter drug metabolism.
* Patients who have received prior therapy with bevacizumab, or related drugs (previous therapy with carboplatin is allowed).
* Inadequately controlled hypertension (defined as systolic blood pressure >150 millimeters of mercury (mmHg) and/or diastolic blood pressure > 100 mmHg) despite antihypertensive medication.
* New York Heart Association (NYHA) Grade II or greater congestive heart failure.
* History of myocardial infarction or unstable angina within 12 months prior to Day 1.
* History of stroke or transient ischemic attack.
* Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1.
* History of hemoptysis (greater than or equal to 1/2 teaspoon of bright red blood per episode) within 1 month prior to Day 1.
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation). (To be eligible, Prothrombin time/international normalized ratio (prothrombin time (PT) international normalized ratio (INR)) should be < 1.4 for patients not on warfarin.)
* Patients receiving full-dose anticoagulants therapy (e.g., warfarin or Low-molecular-weigh (LMW) heparin) and does not meet both of the following criteria:
* No active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices).
* In-range INR (usually between 2 and 3) on a stable dose of oral anticoagulant or on a stable dose of low molecular weight heparin.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 of treatment or anticipation of need for major surgical procedure during the course of the study.
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1.
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1.
* Serious, non-healing wound, active ulcer, or untreated bone fracture.
* Proteinuria as demonstrated by a urine protein:creatinine (UPC) ratio greater than or equal to 1.0 at screening, or Urine dipstick for proteinuria greater than or equal to 2+ (patients discovered to have greater than or equal to 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate less than or equal to 1g of protein in 24 hours to be eligible).
* Known hypersensitivity to any component of bevacizumab.
* Patients has current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, or stable chronic liver disease per investigator assessment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-04-27 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2021-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Camphausen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - Massachusetts General Hospital/Dana Farber, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
We will share coded, linked data in an National Institutes of Health-funded or approved public repository; coded, linked data in another public repository; coded, linked data in Biomedical Translational Research Information System (BTRIS), and identified or coded, linked data with approved outside collaborators under appropriate agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be shared before publication and at the time of publication or shortly thereafter.
Access Criteria: Data will be shared through an National Institutes of Health funded or approved public repository (clinicaltrials.gov); Biomedical Translational Research Information System (BTRIS), and approved outside collaborators under appropriate individual agreements.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-C-0009.html

RESULTS

PARTICIPANT FLOW:
Groups:
- 1/Carboplatin and Bevacizumab for Recurrent Ependymoma: The total duration of treatment will be 6 cycles. After cycle 6, carboplatin should be discontinued, but bevacizumab may be continued at the discretion of the treating physician.
  Carboplatin: Carboplatin will be given on day 1 of each cycle; the carboplatin dose should be calculated using the Calvert formula: Carboplatin dose (mg) = target Area Under the Curve (AUC) x (Creatinine clearance (CrCl) + 25; The total duration of treatment will be 6 cycles. After cycle 6, carboplatin should be discontinued, but bevacizumab may be continued at the discretion of the treating physician
  Bevacizumab: Bevacizumab will be administered on days 1 and 15 of each cycle. Bevacizumab will be administered at a dose of 10 mg/kg; The total duration of treatment will be 6 cycles. After cycle 6, carboplatin should be discontinued, but bevacizumab may be continued at the discretion of the treating physician.
Period: Overall Study
Arm/Group | 1/Carboplatin and Bevacizumab for Recurrent Ependymoma
Started | 35
Completed | 15
Not Completed | 20
Not completed — Switched to alternative treatment | 1
Not completed — Ineligible | 9
Not completed — Withdrawal by Subject | 1
Not completed — Participant chose to be treated in Peru | 1
Not completed — Participant wanting a local endoscopy surgery to remove more tumor | 1
Not completed — Physician Decision | 1
Not completed — Participant decided to pursue other treatment before beginning protocol treatment | 1
Not completed — Disease progression | 4
Not completed — Transferred care before starting new treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | 1/Carboplatin and Bevacizumab for Recurrent Ependymoma
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.497 (16.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 29
  More than one race | 0
  Unknown or Not Reported | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 3
  Not Hispanic | 5
  Unknown | 1
  Missing | 26
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants That Have Progressive Free Survival (PFS) After 1 Year
Description: Percentage of participants that have progressive disease after 1 year. Kaplan-Meier method is used for the analyses of PFS. Progression is a 25% increase in the sum of products of all measurable lesions over smallest sum observed (over baseline if no decrease) using the same techniques as baseline. Clear worsening of any evaluable disease, or appearance of any new lesion/site, clear clinical worsening or failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer).
Time Frame: 1 year
Population: A total of 35 participants were registered, of which 22 were evaluable. 9 participants were screen failures.4 participants withdrew consent prior to starting treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 1/Carboplatin and Bevacizumab for Recurrent Ependymoma
Number analyzed (Participants) | 22
Percentage of participants | 76.4 [52.2 to 89.4]

2. Secondary Outcome: Number of Participants With a (Complete Response (CR) + Partial Response (PR))
Description: Response was measured by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete Response (CR) is complete disappearance of all measurable and evaluable disease. No new lesions. Partial Response (PR) is greater than or equal to 50% decrease under baseline in the sum of products of perpendicular diameters of all measurable lesions.
Time Frame: Up to 6 months and 1 week
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Carboplatin and Bevacizumab for Recurrent Ependymoma
Number analyzed (Participants) | 22
Participants
  Complete Response | 0
  Partial Response | 2

3. Secondary Outcome: Overall Survival (OS)
Description: OS was calculated by the Kaplan Meier methodology. OS is defined as the time from treatment start date until date of death or date last known alive.
Time Frame: The time from treatment start date until date of death or date last known alive, up to 68 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 1/Carboplatin and Bevacizumab for Recurrent Ependymoma
Number analyzed (Participants) | 22
Months | 18.0 [12.2 to NA] — Due to the small sample size, the upper confidence interval (CI) for the Kaplan-Meier curve for OS is never lower than 0.5, for which the median OS correspond to, therefore the upper CI for the median OS does not exist.

4. Secondary Outcome: Mean Core Symptom Severity With Daily Activities Using the MD Anderson Symptom Inventory for Brain Tumors (MDASI-BT)
Description: The MDASI-BT consists of 23 symptoms rated on an 11 point scale (0 - not present, to 10 - as bad as you can imagine) to indicate the presence and severity of the symptom. All participants with at least one valid questionnaire are included in the analyses. We calculated the mean core symptom severity score rated on the scale from 0-not present to 10-as bad as you can imagine at the time of clinical evaluation. Differences of at least 2 points will be classified as the minimum clinically meaningful change in the symptom severity measures. For example, an increase of 2 points or more would mean a moderate improvement, whereas a decrease of 2 points or more would be interpreted as moderate worsening.
Time Frame: Completed at baseline, before a brain or spine magnetic resonance imaging (MRI)/clinical evaluation, and at cycle 2, cycle 4, and cycle 6 (each cycle is 28 days)
Population: 17/22 participants were analyzed because 4 completed the MDASI-SP questionnaires only, and 1 participant completed their baseline assessment 6 days into the first cycle and was not counted.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1/Carboplatin and Bevacizumab for Recurrent Ependymoma
Number analyzed (Participants) | 17
score on a scale
  Baseline | 1.5 (1.8)
  Cycle 2: number analyzed (Participants) | 16
  Cycle 2 | 2.1 (2.1)
  Cycle 4: number analyzed (Participants) | 11
  Cycle 4 | 1.3 (1.1)
  Cycle 6: number analyzed (Participants) | 7
  Cycle 6 | 1.9 (2.0)

5. Secondary Outcome: Mean Core Symptom Severity With Daily Activities Using the MD Anderson Symptom Inventory for Spine Tumors (MDASI-SP) Instrument
Description: The MDASI-SP consists of 23 symptoms rated on an 11 point scale (0 - not present, to 10 - as bad as you can imagine) to indicate the presence and severity of the symptom. All participants with at least one valid questionnaire are included in the analyses. We calculated the mean core symptom severity score rated on the scale from 0-not present to 10-as bad as you can imagine at the time of clinical evaluation. Differences of at least 2 points will be classified as the minimum clinically meaningful change in the symptom severity measures. For example, an increase of 2 points or more would mean a moderate improvement, whereas a decrease of 2 points or more would be interpreted as moderate worsening.
Time Frame: as for outcome 4
Population: 7/22 participants were analyzed because 14 completed the MDASI-BT questionnaires only, and 1 participant completed their baseline assessment 6 days into the first cycle and was not counted.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1/Carboplatin and Bevacizumab for Recurrent Ependymoma
Number analyzed (Participants) | 7
score on a scale
  Baseline: number analyzed (Participants) | 6
  Baseline | 1.4 (0.9)
  Cycle 2 | 2.1 (1.7)
  Cycle 4: number analyzed (Participants) | 5
  Cycle 4 | 2.1 (1.6)
  Cycle 6: number analyzed (Participants) | 1
  Cycle 6 | 1.5 (0)

6. Secondary Outcome: Mean Symptom Interference With Daily Activities Using the MD Anderson Symptom Inventory for Brain Tumors (MDASI-BT)
Description: The MDASI-BT consists of 23 symptoms rated on an 11 point scale (0 - did not interfere, to 10 - interfered completely) to indicate the symptoms that interfere with a participants life in the last 24 hours. All participants with at least one valid questionnaire are included in the analyses. We calculated the mean core symptom interference score rated on the scale from 0- did not interfere, to 10- interfered completely at the time of clinical evaluation. Differences of at least 2 points will be classified as the minimum clinically meaningful change in the symptom interference measures. For example, an increase of 2 points or more would mean a moderate improvement, whereas a decrease of 2 points or more would be interpreted as moderate worsening.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1/Carboplatin and Bevacizumab for Recurrent Ependymoma
Number analyzed (Participants) | 17
score on a scale
  Baseline | 1.6 (2.1)
  Cycle 2: number analyzed (Participants) | 16
  Cycle 2 | 2.1 (2.3)
  Cycle 4: number analyzed (Participants) | 11
  Cycle 4 | 1.7 (1.9)
  Cycle 6: number analyzed (Participants) | 7
  Cycle 6 | 2.5 (2.8)

7. Secondary Outcome: Mean Symptom Interference With Daily Activities Using the MD Anderson Symptom Inventory for Spine Tumors (MDASI-SP) Instrument
Description: The MDASI-SP consists of 23 symptoms rated on an 11 point scale (0 - did not interfere, to 10 - interfered completely) to indicate the symptoms that interfere with a participants life in the last 24 hours. All participants with at least one valid questionnaire are included in the analyses. We calculated the mean core symptom interference score rated on the scale from 0- did not interfere, to 10- interfered completely at the time of clinical evaluation. Differences of at least 2 points will be classified as the minimum clinically meaningful change in the symptom interference measures. For example, an increase of 2 points or more would mean a moderate improvement, whereas a decrease of 2 points or more would be interpreted as moderate worsening.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1/Carboplatin and Bevacizumab for Recurrent Ependymoma
Number analyzed (Participants) | 7
score on a scale
  Baseline: number analyzed (Participants) | 6
  Baseline | 1.7 (1.4)
  Cycle 2 | 3.1 (2.4)
  Cycle 4: number analyzed (Participants) | 5
  Cycle 4 | 4.1 (3.2)
  Cycle 6: number analyzed (Participants) | 1
  Cycle 6 | 4.2 (0)

8. Other Pre Specified Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately, 112 months and 28 days.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Carboplatin and Bevacizumab for Recurrent Ependymoma
Number analyzed (Participants) | 22
Participants | 22

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately, 112 months and 28 days.
Arm/Group | 1/Carboplatin and Bevacizumab for Recurrent Ependymoma
All-Cause Mortality (participants affected / at risk) | 7/35
Serious Adverse Events (participants affected / at risk) | 3/35
Other Adverse Events (participants affected / at risk) | 22/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1/Carboplatin and Bevacizumab for Recurrent Ependymoma (N=35)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2)
Seizure (Nervous system disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1/Carboplatin and Bevacizumab for Recurrent Ependymoma (N=35)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Agitation (Psychiatric disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (5)
Alkaline phosphatase increased (Investigations) | 4 (4)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 8 (35)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (12)
Ataxia (Nervous system disorders) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bloating (Gastrointestinal disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Chills (General disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 7 (7)
Creatinine increased (Investigations) | 3 (7)
Cushingoid (Endocrine disorders) | 1 (1)
Depression (Psychiatric disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Dizziness (Nervous system disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4)
Dysesthesia (Nervous system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Dysphasia (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Eye disorders - Other, Diplopia or double vision (Eye disorders) | 1 (1)
Eye disorders - Other, Peripheral vision (Eye disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Fatigue (General disorders) | 11 (16)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)
Gait disturbance (General disorders) | 3 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 8 (11)
Hematuria (Renal and urinary disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (13)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (16)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 7 (12)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (8)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Investigations - Other, Alanine aminotransferase decreased (Investigations) | 1 (1)
Investigations - Other, specify (Investigations) | 1 (1)
Irregular menstruation (Reproductive system and breast disorders) | 1 (1)
Irritability (General disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 7 (21)
Memory impairment (Nervous system disorders) | 3 (3)
Metabolism and nutrition disorders - Other, Phosphorus count increased (Metabolism and nutrition disorders) | 1 (2)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 3 (3)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 9 (18)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (2)
Nervous system disorders - Other, insomnia (Nervous system disorders) | 1 (1)
Nervous system disorders - Other, left-sided numbness (Nervous system disorders) | 1 (1)
Nervous system disorders - Other, right tongue nymbness (Nervous system disorders) | 1 (1)
Nervous system disorders - Other, neuropathy (Nervous system disorders) | 1 (2)
Neutrophil count decreased (Investigations) | 11 (57)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 2 (3)
Palpitations (Cardiac disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 2 (2)
Periodontal disease (Gastrointestinal disorders) | 1 (1)
Platelet count decreased (Investigations) | 12 (64)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 3 (8)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Renal and urinary disorders - Other, rectal bleeding (Renal and urinary disorders) | 1 (1)
Rhinitis infective (Infections and infestations) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Transient ischemic attacks (Nervous system disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (5)
White blood cell decreased (Investigations) | 11 (45)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2025-07-22): https://cdn.clinicaltrials.gov/large-docs/44/NCT01295944/Prot_SAP_004.pdf
  • Informed Consent Form: Standard Consent (i.e., Clinical Center until 042417) (2017-08-07): https://cdn.clinicaltrials.gov/large-docs/44/NCT01295944/ICF_001.pdf
  • Informed Consent Form: Standard Model Consent (outside sites) (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/44/NCT01295944/ICF_003.pdf